CLINICAL TRIAL: NCT05208346
Title: Acute Effects of Canola Oil Compared With Coconut Oil on Postprandial Metabolism in Women and Men With Increased Risk for Cardiometabolic Diseases
Brief Title: Effects of Canola Oil and Coconut Oil on Postprandial Metabolism in Older Adults With Increased Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: Union for the Promotion of Oil and Protein Plants (UFOP, Germany) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Prof. Dr. Sarah Egert, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 528/191
Record Dates: First submitted 2021-11-23; First posted 2022-01-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome
Keywords: Postprandial metabolic events
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Canola oil high-fat (Experimental): Participants randomized to receive a mixed meal with 50 g canola oil
  Interventions: Dietary Supplement: Mixed meals
- Coconut oil high-fat (Experimental): Participants randomized to receive a mixed meal with 50 g coconut oil
  Interventions: Dietary Supplement: Mixed meals
- Canola oil low-fat (Experimental): Participants randomized to receive a mixed meal with 25 g canola oil
  Interventions: Dietary Supplement: Mixed meals
- Coconut oil low-fat (Experimental): Participants randomized to receive a mixed meal with 25 g coconut oil
  Interventions: Dietary Supplement: Mixed meals

INTERVENTIONS:
Dietary Supplement: Mixed meals — Mixed meals enriched with either 25 or 50 g of canola or coconut oil

SUMMARY:
The aim of this study is to investigate the postprandial effects of fat content and fatty acid composition of mixed meals on parameters associated with cardiometabolic diseases. Therefore, older subjects with increased risk of cardiometabolic diseases consume 4 mixed meals with 25 or 50 g of either canola or coconut oil. In a postprandial period of 6 hours, outcomes associated with cardiometabolic risk (e.g., triglycerides) are analyzed.

DETAILED DESCRIPTION:
In a crossover design, 30 older men and women with increased risk of cardiometabolic diseases consume 4 mixed meals, enriched with either 25 or 50 g canola or coconut oil. During a postprandial period of 6 hours, parameters of lipid metabolism (e.g., plasma triglycerides), glucose metabolism (e.g., plasma glucose, serum insulin), as well as markers of inflammation (e.g., IL-6), vascular system (e.g., pulse wave velocity) and antioxidant system (e.g., trolox equivalent antioxidative capacity) are analyzed. Furthermore, fatty acid profile, neuropsychologic parameters (e.g., attention), subjective feeling of hunger and satiety, and satiety-associated hormones (e.g., ghrelin) are assessed. Each intervention arm will be separated by a washout period of about 14 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 27 - 34,9 kg/m2
* Waist circumference: women ≥ 80 cm, men ≥ 94 cm
* At least two of the following criteria of metabolic syndrome:

Fasting triglycerides in serum: ≥ 150 mg/dl Fasting HDL-Cholesterol in serum: women < 50 mg/dl, men < 40 mg/dl Systolic blood pressure: ≥ 130 mmHg, diastolic blood pressure: ≥ 85 mmHg Fasting glucose in plasma: ≥ 100 mg/dL

Exclusion Criteria:

* Smoking
* Diseases that may impact outcome measures (e.g., thyroid diseases, insulin-dependent diabetes mellitus, impaired renal function, tumors, anemia)
* Intake of immunosuppressives or supplements (e.g., fish oil)
* Participation in another study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Parameters of lipid metabolism in blood I | Postprandial period of 6 hours
  Measurement of triglycerides (mg/dl)
Parameters of lipid metabolism in blood II | Postprandial period of 6 hours
  Measurement of total cholesterol (mg/dl)
Parameters of lipid metabolism in blood III | Postprandial period of 6 hours
  Measurement of LDL cholesterol (mg/dl)
Parameters of lipid metabolism in blood IV | Postprandial period of 6 hours
  Measurement of HDL cholesterol (mg/dl)
Parameters of lipid metabolism in blood VI | Postprandial period of 6 hours
  Measurement of free fatty acids (mmol/L)
Parameters of glucose metabolism in blood I | Postprandial period of 6 hours
  Measurement of glucose (mg/dl)
Parameters of glucose metabolism in blood II | Postprandial period of 6 hours
  Measurement of insulin (nmol/L)

SECONDARY OUTCOMES:
Assessment of hunger and satiety | Postprandial period of 6 hours
  Assessment via visual analogue scales (e.g., 0 = not hungry at all, 10 = very hungry)
Assessment of gut hormones | Postprandial period of 6 hours
  Measurement of gut hormones associated with hunger and satiety in blood (ghrelin in pg/ml; PYY in pg/ml)
Assessment of attention and memory | Postprandial period of 6 hours
  Assessment via validated neuropsychological questionnaires (paper-pencil)
Postprandial endothelial function | Postprandial period of 6 hours
  Assessment via the Vicorder device (e.g., measurement of pulse wave velocity in m/s)
Postprandial inflammation | Postprandial period of 6 hours
  Measurement of parameters of inflammation in blood (e.g., IL-6 in pg/ml)
Antioxidant system | Postprandial period of 6 hours
  Measurement of parameters of antioxidant system in blood (e.g., TEAC in mmol Trolox equivalents/L)
Fatty acid profile | Postprandial period of 6 hours
  Analysis of fatty acid profile in serum (e.g., alpha-linolenic acid in µmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Egert, Prof. Dr., Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany

REFERENCES:
- [Derived] Diekmann C, Schiemann TB, Kienes HF, Wiechmann C, Kopp C, Stoffel-Wagner B, Coenen M, Nemeth R, Wagner M, Egert S. Fat Amount Rather Than Fatty Acid Composition Influences Postprandial Hunger, Satiety and Attention in Men and Women with a Risk Phenotype for Cardiometabolic Diseases: A Randomized Crossover Trial. J Nutr. 2026 Jan;156(1):101232. doi: 10.1016/j.tjnut.2025.11.003. Epub 2025 Nov 11. PMID 41232773